CLINICAL TRIAL: NCT06331039
Title: Investigation of the Effects of Pelvic Floor Muscle Training Combined With Otago Exercises on Symptoms, Balance and Functional Status in Elderly People With UI Living in Nursing Homes
Brief Title: The Effects of Pelvic Floor Muscle Training Combined With Otago Exercises in Elderly People With Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other); Hacettepe University (Other); Dokuz Eylul University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CelalBayarU-5
Record Dates: First submitted 2024-02-05; First posted 2024-03-26 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Urinary Incontinence; Pelvic Floor Muscle Weakness; Muscle Weakness
Keywords: urinary incontinence; pelvic floor muscle training; elektromyography; balance exercises; Otago Exercises
MeSH Terms: conditions — Urinary Incontinence; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFMT+Balance Group (Experimental): PFMT+Otago group was included in the program that includes Otago exercises and pelvic floor muscle training. Otago exercises combined with pelvic floor muscle training will be performed 3 days a week (with a 1-day rest gap between 2 sessions) for 45 minutes per day. Otago exercises consist of strengthening, balance exercises and walking program. Warm-up exercises were performed before each program and cooling exercises were performed at the end of the program. Exercises were performed for 45-60 minutes in each session.
  Interventions: Other: PFMT+Otago
- PFMT Group (Experimental): PFMT group was included in a program that includes pelvic floor muscle training, 3 days a week (with 1 day of rest between 2 sessions) and 45 minutes per day.
  Interventions: Other: PFMT

INTERVENTIONS:
Other: PFMT — PFM exercises were done. Each session were 45 minutes, 2 days a week on a group basis with the physiotherapist, and 1 day a week as a home program, for 12 weeks.
  Arms: PFMT Group
Other: PFMT+Otago — It were done by combining Otago exercises and PFM exercises. Each session were 45 minutes, 2 days a week on a group basis with the physiotherapist, and 1 day a week as a home program, for 12 weeks.
  Arms: PFMT+Balance Group

SUMMARY:
Pelvic floor muscle weakness is one of the most important causes of incontinence. There are many studies supporting that pelvic floor muscle training prevents incontinence and reduces symptom severity, and with A level of evidence, it is among the first in the conservative treatment of incontinence. Functional status and balance problems are common in elderly people with incontinence, and it is known that functional type incontinence is common. Elderly people with incontinence most often fall while trying to get to the toilet. Balance exercises are recommended for falls and balance problems.

The aim of this study is to examine whether pelvic floor muscle training (PFMT) combined with Otago exercises is effective on symptoms, balance and functional status in elderly people with UI living in nursing homes, compared to PFMT alone.

DETAILED DESCRIPTION:
The research was conducted on participants over the age of 65 with urinary incontinence living in a nursing home. After these participants were informed about the content of the study, a signed informed consent form will be obtained. This study is an assessor-blinded, randomized controlled trial. Participants with incontinence aged 65 and over living in a nursig home were randomly assigned to intervention (IG) and control group (CG). The intervention group attended an exercise program that included Otago exercises combined with pelvic floor muscle training (PFMT). The control group was included in the PFMT program with different positions. Duration of exercise for both groups was 45-60 minutes per session three times a week for 12 weeks. Incontinence symptoms and severity (Pelvic Floor Distress Inventory-20, bladder diary), PFM muscle function (superficial electromyography), balance (Berg Balance Scale), functional status (Senior Fitness Test) and fear of falling (Falls Efficacy Scale) was measured at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed the informed volunteer consent form
2. Being 65 years or older
3. Having urinary incontinence
4. Ability to walk unaided and not use any walking aids

Exclusion Criteria:

1. Having severe walking and balance problems
2. Severe cognitive impairment (Mini mental state assessment test score below 23)
3. Having a serious neurological problem
4. Having serious heart diseases
5. Having a genito-urinary infection
6. Having pelvic organ prolapse
7. Six months ago he received medication for incontinence
8. Having had incontinence and abdominal surgery
9. Having metastatic cancer
10. Having any vision problems

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
incontinence symptoms and severity | baseline and week 12 (after intervention)
  SPSS 29 is validated. Pelvic Floor Distress Inventory-20 (PFDI-20) instrument scores were recorded at the baseline and after the intervention. Pelvic Floor Distress Inventory-20 Scale evaluates pelvic organ prolapse, urinary and colorectoanal problems that may develop due to pelvic floor dysfunction, and the degree of complaints about them; It is the short form of the Pelvic Floor Distress Inventory Scale; It consists of 3 subheadings: Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), Urinary Distress Inventory-6 (ÜDI-6) and Colorectoanal Distress Inventory-8 (KRADE-8) and a total of 20 questions. Each subheading score ranges from 0-100, and the total score ranges from 0-300. While the best score for each subheading is 0 and the worst score is 100, the best score in total is 0 and the worst score is 300.
  Change: Week 12- baseline
balance | baseline and week 14 (after intervention)
  SPPS 29 is validated. Berg Balance Scale score will be recorded at baseline and after the intervention. It consists of fourteen items. The proficiency level in the activity for each item is 0; "cannot", 4; It is indicated with 5 points (0-4), "makes it independent and safe". The 14 functional parameters included in Berg Balance Scale. The maximum score that participants can get from the test is 56 and reflects an excellent balance function. (0-20 points; severe fall risk, 21-40 points; moderate fall risk, 41-56; mild fall risk). The fall risk limit for this test is 45 points.
  Change: Week 14- baseline
bladdery diary | baseline and week 12 (after intervention)
  SPPS 29 is validated. Bladdery diary were recorded at the baseline and after the intervention.
  The patient records the type and amount of fluid he/she takes, the frequency of urinary incontinence, the urination volume, the frequency of urination at night, and the situations in which he/she leaks urine, along with the times in a 24-hour voiding diary. It is an objective evaluation method used to determine the type and degree of incontinence.
  Change: Week 12- baseline
Senior fitness test- functional performance-30-second chair stand test | baseline and week 12 (after intervention)
  SPPS 29 is validated. 30-second chair stand test score were recorded at the baseline and after the intervention.
  The participant was asked to sit in the middle part of a 43.18 cm (12in) high chair with his back upright, feet on the ground and arms crossed in front of his chest (right hand on the left shoulder, left hand on the right shoulder). While in this position, the participant starts the test with the start command and takes off as fully as he can during 30 seconds. The number of complete takes off during 30 seconds determines the score.A score of less than 10 in 30 seconds indicates lower extremity muscle weakness.
  Change: Week 12- baseline.
Senior fitness test- functional performance-Eight (2.45m) Food Up and Go Test | baseline and week 12 (after intervention)
  SPPS 29 is validated.For the test, which is used to evaluate functional mobility and dynamic balance in elderly participants, the participants was seated in a chair with a backrest and armrests, with his back and arms supported. After the command to "get up" was given to the patient, he was asked to walk at his normal speed to an object placed 2.45 m away from the chair, and then turn around the object and walk back. The period started when the patient was commanded to "get up" and was stopped when he/she sat on the chair.
  Change: Week 12- baseline.
Senior fitness test- functional performance-Chair Sit and Reach Test | baseline and week 12 (after intervention)
  SPSS 29 is validated.This test, is used especially to determine the flexibility of the hamstring muscle group. The participant was seated on a 43.18 cm high chair leaning against a wall or a solid place, with the junction of the thigh and hip bones in front of the chair. The participant was allowed to extend one foot forward, in full extension, with the heel on the ground and the ankle at approximately 90 degrees, leaving it to the participant's own choice (right or left). The participant was told to stretch his body forward with both hands, without bending his extended knee, and to reach towards his toe without pushing the pain limit. Participant; If the fingertips do not touch the tip of the foot, the distance between them, in centimeters (-), is the participant's; If the fingertips of the middle hand touch the tip of the foot, zero (0) is given to the participant.
Senior fitness test- functional performance-Two Minutes Step Test | baseline and week 12 (after intervention)
  SPPS 29 is validated. In order to perform the test, the participant stands in an upright position; The distance from the front protrusion of the hip bone (iliac crest) to the midpoint of the kneecap (patella) was marked and the midpoint of the distance between these two bones was determined. The participant's step height was determined by marking the height of this determined point from the ground. In order to determine whether the step height reached the target height, a strip was drawn at the determined height or the target height was marked on the wall and it was checked whether the participant's step height (knee height) reached the target height. The participant was made to step where both knees were, reaching the specified height for 2 minutes. At the end of 2 minutes, the total number of right steps taken correctly was recorded.
  Change: Week 12-baseline
Muscle Function- Pelvic floor muscles-Superficial electromyography (EMG) | baseline and week 12 (after intervention).
  SPPS 29 is validated.EMG measurement; It was used to record the bioelectrical activity generated by superficial PFM. In the research, NeuroTrac MyoPlus 4 PRO type EMG device was used. Superficial PFM EMG activities were evaluated using disposable, superficial, self-adhesive, silver-silver chloride (Ag/AgCl) electrodes. The diameter of the circular adhesive electrodes was 3.2 cm. The skin area where the superficial electrodes would be attached was cleaned with an alcohol swab to reduce skin impedance. Superficial electrodes were then placed on the muscles parallel to the muscle fibers: superficial PFM- on both sides of the perineal body. The monopolar reference electrode was placed on the right spina iliac anterior superior (SIAS) to eliminate external signals from outside.
Fear of falling-Fall Efficacy Scale (FES) | baseline and week 12 (after intervention).
  SPPS 29 is validated.The first version of the Falls Efficacy Scale (FES) was developed by Tinetti and colleagues in the form of 10 questions covering simple daily living activities to evaluate the fear of falling in the elderly population. It enables the detection and evaluation of the activities that cause fear in people. The Fall Activity Scale-International, which is frequently used today, was developed by Yardley et al.by modifying and preserving the 10 items in the original scale and adding 6 new items. According to this index, as the score increases, the fear of falling increases (scale score between 0-100).
  Change: Week 12-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Özge ÇELİKER TOSUN, Assoc. Prof., Study Director — Dokuz Eylul University
Locations (1):
- Melda BAŞER SEÇER, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data is saved on my hard disk, I can share it if desired.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: five year
Access Criteria: If it is necessary

REFERENCES:
- [Derived] Baser Secer M, Celiker Tosun O, Akbayrak T, Ilcin N, Tosun G. Does combining two evidence-based exercise programs in elderly people with incontinence have a triple effect on incontinence symptoms, balance and functional status? Int Urol Nephrol. 2025 Jan;57(1):79-91. doi: 10.1007/s11255-024-04177-4. Epub 2024 Aug 1. PMID 39090517